CLINICAL TRIAL: NCT06101459
Title: A Study About Association Between Microbiome, Metabolome and Clinical Characteristics in COPD Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Asan Medical Center (Other)
Collaborators: Seoul National University College of Medicine (Unknown); HEM Pharma Inc. (Industry)
Responsible Party: Principal Investigator, Sei Won Lee, Professor, Asan Medical Center
Other Study IDs: 2023-1049
Record Dates: First submitted 2023-10-19; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Microbiome; Metabolome; Smoking history
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Fecal sample: the investigators will collect fecal sample (≥ 10g) and divided them into stool sample collection kit and OMNIgene GUT OMR-200 Kit (DNA Genotek, Canada).
  Sputum sample: the investigators will collect induced sputum sample from each subject. Induction with hypertonic saline (3%) will be performed.
  Blood sample: the investigators will retrieve 5cc blood sample from each patient. Blood samples will be centrifuged and stored as plasma and peripheral blood mononuclear cells, respectively.
  All samples will be freeze-dried for 24 hours using a benchtop manifold freeze drier and stored at -80°C until analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COPD patient with significant smoking history: Patients with following conditions
  1. smoking history more than 30 pack*year
  2. FEV1/FVC ratio <0.7
  3. No acute exacerbation history within 3 months
- COPD patient without significant smoking history: Patients with following conditions
  1. smoking history less than 0.5 pack*year
  2. FEV1/FVC ratio <0.7
  3. No acute exacerbation history within 3 months
- Healthy smoker: Patients with following conditions
  1. smoking history more than 30 pack*year
  2. FEV1/FVC ratio ≥0.7
  3. No current use of medication for any chronic respiratory disease

SUMMARY:
The goal of this observational registry study is to compare characteristics of gut and sputum microbiome and metabolome among COPD patients with significant smoking history, COPD patients without significant smoking history and healthy smoker. Additionally, the investigators investigate the difference of blood metabolites and peripheral blood mononuclear cells level among groups.

The main questions it aims to answer are:

* Are there significant difference in fecal or sputum microbiome and metabolome between COPD patients and healthy smoker?
* Are there any distinct characteristics in microbiome and metabolome in COPD with COPD patients with significant smoking history, COPD patients without significant smoking history compared with healthy smoker?
* Are there any difference in blood metabolites and peripheral blood mononuclear cells levels among patients with significant smoking history, COPD patients without significant smoking history and healthy smoker
* Might distinct characteristics of microbiome and metabolites in COPD patients be related to worse clinical outcomes in COPD patients?

ELIGIBILITY:
Inclusion Criteria:

* COPD Patients, defined by FEV1/FVC <0.7, who

  * agree with informed consent
  * have no history of acute exacerbation within 3 months
* Healthy smoker without airflow limitation, defined by FEV1/FVC ≥0.7, who

  * have smoking history with at least 30 pack-year
  * agree with informed consent
  * do not use medication for chronic respiratory disease

Exclusion Criteria:

* Withdrawal of informed consent
* History of acute exacerbation or antibiotics use within 3 months
* Difficulty to collect adequate stool, sputum and blood samples

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. COPD patients with significant smoking history
     * FEV1/FVC <0.7 in spirometry
     * Smoking history at least 30 pack-year
  2. COPD patients without significant smoking history
     * FEV1/FVC <0.7 in spirometry
     * No smoking history or smoking history at less than 0.5 pack-year
  3. Healthy smoker
     * FEV1/FVC ≥0.7 in spirometry
     * Smoking history at least 30 pack-year
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Shannon diversity index | At enrollment
  the investigators will compare alpha diversity and community similarity among groups by using the Shannon diversity index.
Simpson index | At enrollment
  the investigators will compare alpha diversity and community similarity among groups by using the Simpson index.
Principal component analysis | At enrollment
  the investigators will compare beta diversity and community similarity among groups by using the principal component analysis.
Microbiome composition by metagenomic analysis | At enrollment
  The composition of microbiome will be presented as bar graph.
Peripheral blood mononuclear cells level | At enrollment
  the investigators will compare the Peripheral blood mononuclear cells level among groups
Acetic acid level | At enrollment
  the investigators will compare the acetic acid level among groups
Propionic acid level | At enrollment
  the investigators will compare the Propionic acid level among groups
Isobutyric acid level | At enrollment
  the investigators will compare the Isobutyric acid level among groups
Butyric acid level | At enrollment
  the investigators will compare the butyric acid level among groups
Isovaleric acid level | At enrollment
  the investigators will compare the Isovaleric acid level among groups
Valeric acid level | At enrollment
  the investigators will compare the valeric acid level among groups
dimethylglycine level | At enrollment
  the investigators will compare the dimethylglycine level among groups
secondary bile acid level | At enrollment
  the investigators will compare the secondary bile acid level among groups

SECONDARY OUTCOMES:
Difference of microbiome according to Exacerbation | within 1 year after enrollment
  the investigators will investigate the baseline difference of microbiome between COPD patients with moderate to severe exacerbation and COPD patients without moderate to severe exacerbation
Difference of metabolome according to Exacerbation | within 1 year after enrollment
  the investigators will investigate the baseline difference of metabolome between COPD patients with moderate to severe exacerbation and COPD patients without moderate to severe exacerbation
Difference of microbiome according to death | within 1 year after enrollment
  the investigators will investigate the baseline difference of microbiome between COPD patients with death and COPD patients without death
Difference of metabolome according to death | within 1 year after enrollment
  the investigators will investigate the baseline difference of metabolome between COPD patients with death and COPD patients without death